CLINICAL TRIAL: NCT05313295
Title: Effects of the Physical Therapy Treatment on Children and Adolescents With Chronic and Neurological Pathologies Affecting Their Sensorimotor Abilities.
Brief Title: Physical Therapy Treatment on Children and Adolescents With Neurological Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Sánchez Joya, Associate Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FiNeuro
Record Dates: First submitted 2022-02-27; First posted 2022-04-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Neurologic Disorder; Duchenne; Pediatric Disorder; Sensorimotor Disorder Nos
Keywords: Childhood; Neurologic disorder; Duchenne
MeSH Terms: conditions — Nervous System Diseases; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Physiotherapy (Experimental): Two days a week of physical therapy (mobilizations, manual therapy, stretching, respiratory techniques) + 3 hours extra of home-based physiotherapy (stretching, active mobilizations)
  Interventions: Other: Home-based physiotherapy
- Usual physiotherapy (Active Comparator): Two days a week of physical therapy (mobilizations, manual therapy, stretching, respiratory techniques)
  Interventions: Other: Usual Physiotherapy

INTERVENTIONS:
Other: Home-based physiotherapy — Manual Therapy, passive and active mobilizations, stretching, respiratory techniques
  Arms: Home-based Physiotherapy
Other: Usual Physiotherapy — Usual care provided for the management of neurological disorders in children
  Arms: Usual physiotherapy

SUMMARY:
To evaluate the positive effects of a home-based physical therapy intervention added to the usual physical therapy programs performed in children with neurological pathologies that induce sensorimotor impairments that affect their quality of life and the importance of the implications of their families in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents agree to include their children on the study
* Affiliated to the Duchenne Parents Project Association (Spain)
* Between 3-18 years old

Exclusion Criteria:

* Other pathological conditions
* Parents refuse the participation on the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure | One Year
  Measurement scale for motor function applied to neuromuscular diseases (MFM): It was created in France in order to perform a better evaluation of global motor function in patients with Duchenne's muscular dystrophy (DMD), both for ambulatory and non-ambulatory patients. It has two versions, MFM 20 for children under 6 years of age and MFM 32 for children over 6 years of age. The scale considers three dimensions: (D1) standing station and transfers; (D2) axial and proximal motor skills and (D3) distal motor skills. The sum of the three results in a global percentage that provides an updated overview of the patient's functional diagnosis. (Trundell et al., 2020)

SECONDARY OUTCOMES:
Brooke Upper Extremity Scale | One Year
  It is a scale of levels from 1 to 5 for the motor functional classification of the upper limbs. (Brooke et al., 1989) It is graded according to the motor ability of the child evaluated in the following categories: (1) bring the arms towards the ceiling (2) raises arms above head but bends elbows (3) cannot raise hands above head, but can bring glass of water to mouth (4) holds pen or picks up coin and ( 5) It does not have any useful function with the hand. The lower the score, the better the upper extremity motor function. (Mayhew et al., 2013) In addition, this scale is frequently used in the DMD population and its intraclass correlation coefficient (ICC) is .99 .(Lue et al., 2006)
Vignos Scale | One Year
  It is a functional classification that scores from 1 to 10, where the highest number represents the most intense progressive condition of DMD reflected in the patient's ambulation. The possible categories are: (1) walks and climbs stairs without assistance (2) walks and climbs stairs with assistance or handrails (3) walks and climbs stairs slowly with the assistance of handrails (4) walks without assistance and gets up from a chair but does not climb stairs (5) walks without assistance but cannot get up from a chair or climb stairs (6) walks only with the aid of long orthoses (7) walks with long orthoses but needs help to maintain balance (8) stands upright with orthoses but unable to walk or with assistance, (9) in a wheelchair and (10) confined to bed.(Fernandes et al., 2014; Martini et al., 2015)
Timed Up and Go Test | One Year
  Determines the patient's risk of falling. The test is performed under a stopwatch, asking the patient to get up from a chair (with or without support), stand up, walk 3 meters, turn around and come back to sit on the chair again. If the patient takes more than 20 seconds to perform, they have a high risk of falling; and between 10 and 20 seconds will indicate fragility. (Alkan et al., 2017)
Six Minutes Walk Distance | One Year
  It consists of quantifying in meters the distance traveled in 6 minutes by the patient. The more meters walked, the less impairment.(Mcdonald et al., 2013) Individualized periodic assessment of 6 Minutes Walking Distance (6MWD) is the most widely accepted primary clinical endpoint in Duchenne's muscular dystrophy (DMD) clinical trials(Goemans et al., 2016); and provides a better prognosis than those based solely on age. After analyzing its test-retest reliability in DMD, its ICC is 0.92. (Mcdonald et al., 2013)

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Sánchez-Joya, PhD, Study Chair — Universidad de Almeria
Locations (1):
- María del Mar Sánchez-Joya, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: SAP
Time Frame: Data will become available for one year once the study is finished
Access Criteria: Reasonable request to reproduce the intervention performed on this study

REFERENCES:
- [Background] Alemdaroglu I, Karaduman A, Yilmaz OT, Topaloglu H. Different types of upper extremity exercise training in Duchenne muscular dystrophy: effects on functional performance, strength, endurance, and ambulation. Muscle Nerve. 2015 May;51(5):697-705. doi: 10.1002/mus.24451. Epub 2015 Mar 5. PMID 25196721
- [Background] Alkan H, Mutlu A, Firat T, Bulut N, Karaduman AA, Yilmaz OT. Effects of functional level on balance in children with Duchenne Muscular Dystrophy. Eur J Paediatr Neurol. 2017 Jul;21(4):635-638. doi: 10.1016/j.ejpn.2017.02.005. Epub 2017 Feb 20. PMID 28259452
- [Background] Hind D, Parkin J, Whitworth V, Rex S, Young T, Hampson L, Sheehan J, Maguire C, Cantrill H, Scott E, Epps H, Main M, Geary M, McMurchie H, Pallant L, Woods D, Freeman J, Lee E, Eagle M, Willis T, Muntoni F, Baxter P. Aquatic therapy for children with Duchenne muscular dystrophy: a pilot feasibility randomised controlled trial and mixed-methods process evaluation. Health Technol Assess. 2017 May;21(27):1-120. doi: 10.3310/hta21270. PMID 28627356
- [Background] Goemans N, Vanden Hauwe M, Signorovitch J, Swallow E, Song J; Collaborative Trajectory Analysis Project (cTAP). Individualized Prediction of Changes in 6-Minute Walk Distance for Patients with Duchenne Muscular Dystrophy. PLoS One. 2016 Oct 13;11(10):e0164684. doi: 10.1371/journal.pone.0164684. eCollection 2016. PMID 27737016
- [Background] Jansen M, van Alfen N, Geurts AC, de Groot IJ. Assisted bicycle training delays functional deterioration in boys with Duchenne muscular dystrophy: the randomized controlled trial "no use is disuse". Neurorehabil Neural Repair. 2013 Nov-Dec;27(9):816-27. doi: 10.1177/1545968313496326. Epub 2013 Jul 24. PMID 23884013